CLINICAL TRIAL: NCT01681316
Title: A Randomized, Multi-center, Double-blind, Placebo-controlled Trial of Danhong Injection in the Treatment of Chronic Stable Angina
Brief Title: Danhong Injection in the Treatment of Chronic Stable Angina
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: China Food and Drug Administration (Other Government)
Responsible Party: Principal Investigator, Zhong Wang, Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DH20120703
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Stable Angina
Keywords: Chronic Stable Angina; Randomized Controlled Trial; Traditional Chinese Medicine
MeSH Terms: conditions — Angina, Stable | interventions — danhong

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Danhong injection (Experimental): Based on the standard medical care, 40ml of Danhong injection, added into 250ml of 0.9% saline, given by continuous IV infusion at 2.5ml/min within 2 hours.
  Interventions: Drug: Danhong injection; Other: Standard medical care
- Placebo (Placebo Comparator): Based on the standard medical care, placebo was 40ml of 0.9% saline, added into 250ml of 0.9% saline, given by continuous IV infusion at 2.5ml/min within 2 hours.
  Interventions: Other: Standard medical care; Drug: Placebo

INTERVENTIONS:
Drug: Danhong injection — A kind of injection made from two kind of Chinese herbs: salvia miltiorrhiza and safflower
  Arms: Danhong injection
Other: Standard medical care — Standard medical care is in accordance with China Guideline for the diagnosis and treatment of Chronic Stable Angina (2007).
Drug: Placebo — 0.9% saline added into 250ml 0.9% saline by an independent research nurse, sealed with brown bag in order to make the investigators and patients blinded, using brown infusion tube for infusion.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of Danhong Injection on the relief of angina with the use of the Seattle Angina Questionnaire among patients with stable angina patients

ELIGIBILITY:
Inclusion Criteria:

* Female or male inpatients.
* Age: 18 - 70 years.
* Patients with clinical diagnosis of chronic stable angina and must meet one of the following conditions:1）Patients who have a history of myocardial infarction and ST-T changes;2）Stenosis of more than 50% in at least one major epicardial coronary artery shown by Coronary Angiograph or CT Angiography; 3）Patients with coronary heart disease were determined by radionuclide angiocardiography.
* Clinical diagnosis of "Xueyu Zheng" (Blood Stasis Syndrome) as the scores of Chinese medicine symptoms scales of "Xueyu Zheng" in angina ≥ 15. The Chinese medicine symptoms scales of "Xueyu Zheng" is defined as following (1)chest pain-10, (2)chest distress-10, (3) palpitation-5, (4)purple or dark lip-5, (5) purple or dark tongue-5, (6) unsmooth pulse-5.
* Patients with moderate angina pectoris (The definition of "moderate angina pectoris " is in accordance with the Canadian Cardiovascular Society (CCS) grading of angina pectoris,which be classified to II or III.
* Patient is willing to participate voluntarily and to sign a written patient informed consent.

Exclusion Criteria:

* Woman with pregnancy, lactation or positive result of pregnancy test, or woman who is under menstrual period.
* Woman who disagree with contraception during treatment period
* Patients with severe complications that would make the condition more complicated assessed by the investigator, including liver or renal dysfunction, severe cardiopulmonary dysfunction, pulmonary hypertension, chronic obstructive pulmonary disease, a history of epilepsy or cerebral hemorrhage .
* Patients who were angina-free during the run-in period without taking any drug.
* Patients with myocardial infarction or Canadian Cardiovascular Society (CCS) grading of angina pectoris class IV within the preceding 3 months
* Patients with chest pain caused by other disease (e.g., acute myocardial infarction，severe neurosis，menopausal syndrome，hyperthyroidism).
* Patients with history of drug-induced bleeding or history of bleeding caused by warfarin.
* Patients with history of hematopoietic system diseases.
* Patients who had surgery within the past 4 weeks and have hemorrhagic tendency.
* Patients who is participating in other trials or has been participated in other trials in recent 3 months.
* Patients with history of allergy or suspected allergic to the drug.
* Patients who were suspected addicted into alcohol or drug abuse in the past 2 years.
* Patients with mental disorder.
* Patients who were unable to participate in the study as judged by investigator.
* Patients who were family members or relatives of the research center staffs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2012-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in each treatment group who had clinically significant change as defined by the angina-frequency score on the Seattle Angina Questionnaire at day 30 | Day 30
  Seattle Angina Questionnaire, a 19-item questionnaire that quantifies physical limitations due to angina, any recent change in the severity of angina, the frequency of angina, satisfaction with treatment, and quality of life. Scores range from 0 to 100; higher scores indicate better health status.With a score of 20 or more on the angina-frequency scale indicating that the patient was clinically significant change.

SECONDARY OUTCOMES:
Total score of symptoms questionnaire of TCM | Day 0, Day 7, Day 14, Day 30, Day 60, Day 90
  The symptoms questionnaire of TCM consists of 6 symptoms that described in traditional Chinese medicine, including chest pain, chest distress, palpitation, dark-purple lip, dark-purple tongue and unsmooth pulse. Each symptom was assessed by the Visual Analogue Scale（VAS），where a higher score meant higher severity.
The proportion of patients in each treatment group who had clinically significant changes in the other four Seattle Angina Questionnaire scales （The physical limitation, angina stability, treatment satisfaction, and quality of life） | Day 0, Day 7, Day 14, Day 30, Day 60, Day 90
  We defined clinical significant changes as a difference of 8 points or more on the physical-limitation scale, 25 or more on the angina-stability scale, 12 or more on the treatment-satisfaction scale, or 16 or more on the quality-of-life scale.
The frequency of anginal attack every week | Day-7 (if exist), Day 0, Day 7, Day 14, Day 30, Day 60, Day 90
  The frequency of anginal attack was recorded by the patients with the use of the diary cards which will be collected from the run-in period (Day -7) to the end of follow-up (Day 90).
Canadian Cardiovascular Society (CCS) grading of angina pectoris | Day 0, Day 7, Day 14, Day 30, Day 60, Day 90
Consumption of Short-acting Nitrates | Day -7( if exist), Day 0, Day 7, Day 14, Day 30, Day 60, Day 90
Change in the electrocardiogram (EKG) | Day 0, Day 7, Day 14, Day 30, Day 60, Day 90
Changes in the Serum Lipid, the high-sensitivity C-Reactive Protein(hs-CRP) and the Platelet Aggregation Rate | Day 0, Day 14
Incidence of new-onset major vascular events in 90 days | Day 90
  Major adverse vascular events include ischemic stroke, hemorrhagic stroke, TIA, myocardial infarction and vascular-related death.
Overall mortality in 90 days | Day 90
Incidence of severe hemorrhages in 90 days | Day 90
  The definition of "Severe hemorrhages" is in accordance with the GUSTO bleeding criteria, including fatal intracranial hemorrhage (ICH), symptomatic intracerebral hemorrhage (sICH) or which could result in substantial hemodynamic compromise requiring treatment.
Incidence of moderate hemorrhages in 90 days | Day 90
  The definition of "moderate hemorrhages" is in accordance with the GUSTO bleeding criteria, which requires blood transfusion but not results in hemodynamic compromise.
Documentation of adverse events (AEs) and serious AEs | 90 days

OTHER OUTCOMES:
The profiles of micro-RNA in 60 patients selected from certain centers | Day 0, Day 14, Day 90
The profiles of mRNA in 60 patients selected from certain centers | Day 0, Day 14, Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, Professor, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Yun-dai Chen, Professor, Principal Investigator — Chinese PLA General Hospital(301 Hospital); Yong-yan Wang, Professor, Study Chair — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Xiao-xi Du, Professor, Study Director — China Food and Drug Administration
Locations (31):
- China (31):
  - Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Xuan Wu Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Dongfang Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital(301 Hospital), Beijing, Beijing Municipality
  - Chongqing Traditional Chinese Medicine Hopital, Chongqing, Chongqing Municipality
  - The Third People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Heilongjiang University of Traditional Chinese Medicine, Harbin, Heilongjiang
  - The First Affiliated Hospital of Heilongjiang University of Traditional Chinese Medicine, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of T.C.M., Zhengzhou, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Provincial Hospital of T.C.M., Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - The First Hospital of Changsha, Changsha, Hunan
  - The Second Affiliated Hospital to Hunan University of Chinese Medicine, Changsha, Hunan
  - Jilin Province People's Hospital, Changchun, Jilin
  - The Affiliated Hospital to Changchun University of Chinese Medicine, Changchun, Jilin
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital to Shanxi Medical University, Taiyuan, Shanxi
  - Affiliated Hospital of Shanxi University of Chinese Medicine, Xianyang, Shanxi
  - Xi'an City Hospital of T.C.M., Xi’an, Shanxi
  - Shanxi Province Hosptial of T.C.M., Xi’an, Shanxi
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - Chengdu Sencond People's Hospital, Chengdu, Sichuan
  - Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Xin Hua Hospital of Zhejiang Province, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Guan S, Yu YN, Li B, Gu H, Chen L, Wang N, Wang B, Liu X, Liu J, Wang Z. Discovery of Drug-Responsive Phenomic Alteration-Related Driver Genes in the Treatment of Coronary Heart Disease. Pharmgenomics Pers Med. 2023 Mar 15;16:201-217. doi: 10.2147/PGPM.S398522. eCollection 2023. PMID 36945217
- [Derived] Liu J, Li DD, Dong W, Liu YQ, Wu Y, Tang DX, Zhang FC, Qiu M, Hua Q, He JY, Li J, Du B, Du TH, Niu LL, Jiang XJ, Cui B, Chen JB, Wang YG, Wang HR, Yu Q, He J, Mao YL, Bin XF, Deng Y, Tian YD, Han QH, Liu DJ, Duan LQ, Zhao MJ, Zhang CY, Dai HY, Li ZH, Xiao Y, Hu YZ, Huang XY, Xing K, Jiang X, Liu CF, An J, Li FC, Tao T, Jiang JF, Yang Y, Dong YR, Zhang L, Fu G, Li Y, Huang SW, Dou LP, Sun LJ, Zhao YQ, Li J, Xia Y, Liu J, Liu F, He WJ, Li Y, Tan JC, Lin Y, Zhou YB, Yang JF, Ma GQ, Chen HJ, Liu HP, Liu ZW, Liu JX, Luo XJ, Bin XH, Yu YN, Dang HX, Li B, Teng F, Qiao WM, Zhu XL, Chen BW, Chen QG, Shen CT, Wang YY, Chen YD, Wang Z. Detection of an anti-angina therapeutic module in the effective population treated by a multi-target drug Danhong injection: a randomized trial. Signal Transduct Target Ther. 2021 Sep 1;6(1):329. doi: 10.1038/s41392-021-00741-x. PMID 34471087
- [Derived] Wang PQ, Li DD, Dong W, Liu J, Yu YN, Shen CT, Chen QG, Chen BW, Chen YD, Wang Z. Danhong injection in the treatment of chronic stable angina: study protocol for a randomized controlled trial. Trials. 2015 Oct 21;16:474. doi: 10.1186/s13063-015-0998-1. PMID 26489511